CLINICAL TRIAL: NCT00426608
Title: Placebo-Controlled, Randomized, Blinded, Double-Dummy, Crossover Study to Investigate the Attenuation of ACTH Activation Induced by Metyrapone With a Single Dose of GSK561679 or Alprazolam in Healthy Volunteers
Brief Title: To Investigate Effects GSK561679 on Part of the Body's System That Controls the Balance of Many of the Hormones.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Diagnostic
Other Study IDs: CRS105511
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: HPA axis,; Healthy volunteers; hormones,; GSK561679,; cortisol,
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Metyrapone; Alprazolam; NBI 77860

ARMS (5):
- Session 1 (Experimental): Subjects will be randomized to receive Dose 1 of Metyrapone 0.04 gram per kilogram (g/kg) and Dose 2 of AEBCD sequence. In AEBCD sequence A is placebo, E Alprazolam, B GSK6561679 10 milligram (mg), C GSK6561679 50 mg and D GSK6561679 400 mg. Wash-out period will be of 7 days.
  Interventions: Drug: metyrapone; Drug: alprazolam; Drug: placebo; Drug: GSK561679
- Session 2 (Experimental): Subjects will be randomized to receive Dose 1 of Metyrapone 0.04 g/kg and Dose 2 of BACED sequence. In BACED sequence B is GSK6561679 10 mg, A placebo, C GSK6561679 50 mg, E Alprazolam, and D GSK6561679 400 mg. Wash-out period will be of 7 days.
  Interventions: Drug: metyrapone; Drug: alprazolam; Drug: placebo; Drug: GSK561679
- Session 3 (Experimental): Subjects will be randomized to receive Dose 1 of Metyrapone 0.04 g/kg and Dose 2 of CBEAD sequence. In CBEAD sequence C is GSK6561679 50 mg, B GSK6561679 10 mg, E Alprazolam, A placebo, and D GSK6561679 400 mg. Wash-out period will be of 7 days.
  Interventions: Drug: metyrapone; Drug: alprazolam; Drug: placebo; Drug: GSK561679
- Session 4 (Experimental): Subjects will be randomized to receive Dose 1 of Metyrapone 0.04 g/kg and Dose 2 of ECABD sequence. In ECABD sequence E is Alprazolam, C is GSK6561679 50 mg, A placebo, B GSK6561679 10 mg and D GSK6561679 400 mg. Wash-out period will be of 7 days.
  Interventions: Drug: metyrapone; Drug: alprazolam; Drug: placebo; Drug: GSK561679
- Session 5 (Experimental): Subjects will be randomized to receive Dose 1 of Metyrapone 0.04 g/kg and Dose 2 of GSK561679 400 mg and alprazopam placebo. Wash-out period will be of 7 days.
  Interventions: Drug: metyrapone; Drug: alprazolam; Drug: placebo; Drug: GSK561679

INTERVENTIONS:
Drug: metyrapone — Metyrapone will be available as 250 mg dose capsule.
Drug: alprazolam — Alprazolam capsules will be available with dose strength of 0.25mg
Drug: placebo — GSK561679 placebo tablets visually match the active GSK561679 tablets. Placebo to match Alprazolam is a hard gelatine capsule that visually matches active Alprazolam capsules.
Drug: GSK561679 — GSK561679 tablets will be available with dose strength of 50, 10 and 200 mg.
  Other Names: Single dose of GSK561679; Single dose of metyrapone; Single dose of placebo; Single dose of alprazolam

SUMMARY:
A study to investigate the effects GSK561679 on part of the body's system that controls the balance of many of the hormones (including cortisol).

ELIGIBILITY:
Inclusion:

* Healthy male subjects
* non-smoker
* normal ECG

Exclusion:

* shift workers
* vegetarians
* persons who travel distances
* persons participating in a psychology or psychiatry course

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10-06 (Actual); Primary Completion 2007-01-08 (Actual); Study Completion 2007-01-08 (Actual)

PRIMARY OUTCOMES:
Blood levels of ACTH: over 24 hours | Over 24 hours

SECONDARY OUTCOMES:
Blood levels of GSK561679, metyrapone, alprazolam, cortisol: over 24 hours Questionnaires: each visit Safety (ECG/vital signs/Adverse Events/ laboratory): over 24 hours | Over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study CRS105511 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/CRS105511?search=study&search_terms=CRS105511#rs